CLINICAL TRIAL: NCT01629199
Title: The Clinical Trial for Evaluation of Efficacy and Safety of rhEGF(Recombinant Human Epidermal Growth Factor) in Diabetic Foot Ulcer Patients With Uncontrolled Diabetes Mellitus.
Brief Title: Efficacy and Safety of rhEGF in Diabetic Foot Ulcer Patients With Uncontrolled Diabetic Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW-EGF011P
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Diabetic Foot Ulcer Patients With Uncontrolled Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- rhEGF(recombinant human Epidermal Growth Factor) (Experimental): BID
  Interventions: Drug: rhEGF(recombinant human Epidermal Growth Factor)
- placebo (Placebo Comparator): BID
  Interventions: Drug: placebo of rhEGF(recombinant human Epidermal Growth Factor)

INTERVENTIONS:
Drug: rhEGF(recombinant human Epidermal Growth Factor)
  Arms: rhEGF(recombinant human Epidermal Growth Factor)
Drug: placebo of rhEGF(recombinant human Epidermal Growth Factor)
  Arms: placebo

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and efficacy of rhEGF (recombinant human Epidermal Growth Factor) in diabetic foot ulcer patients with uncontrolled diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
At 12 weeks, wound closure rate of diabetic foot ulcers | 12 weeks from the start day of treatment (But, the study can be finished before 12 weeks)

SECONDARY OUTCOMES:
Time to reach complete wound closure | 12weeks
average size reduction of diabetic ulcer | 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- College of Medicine, Yonsei University, Seoul, South Korea